CLINICAL TRIAL: NCT05149664
Title: A Non-significant Risk Clinical Study to Assess Changes in Perfusion Resulting From Application of the VibratoSleeve, a Therapeutic Ultrasound (TUS) Phased Array, for Patients With Peripheral Arterial Disease (PAD)
Brief Title: A Non-significant Risk Clinical Study: Changes in Perfusion After Therapeutic Ultrasound in Patients With PAD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vibrato Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S21-002 (Prelude Study)
Record Dates: First submitted 2021-10-21; First posted 2021-12-08 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Peripheral Arterial Disease (PAD)
Keywords: Therapeutic Ultrasound (TUS)
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Ultrasonic Therapy

STUDY DESIGN:
Intervention Model Description: Prospective, single arm, open-label design of the VibratoSleeve TUS device.
Masking Description: N/R
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- VibratoSleeve TUS (Experimental): Subjects will receive 30 TUS treatments, each one lasting 90 minutes on the calf of a leg with peripheral arterial disease.
  Interventions: Device: Therapeutic ultrasound (TUS)

INTERVENTIONS:
Device: Therapeutic ultrasound (TUS) — As described elsewhere, a sleeve is wrapped around the subject's targeted calf such that the inner lining with attached transducers are positioned around the calf muscle, with a gel-skin interface. The ultrasound energy is transmitted from these transducers to the deeper layers of the muscle.

SUMMARY:
All evaluable subjects will receive VibratoSleeve therapeutic ultrasound (TUS) treatments. The device will be programmed to deliver TUS at a pre-determined level. Three different acoustic intensity levels will be tested during the first three treatment visits (one at each visit day). The most effective treatment that is comfortable to a subject will be prescribed for the remaining treatment sessions. Treatment time will be 90 minutes per session, one session per day. Thirty treatment sessions will be performed over a 45-day period.

Subjects will appear for on-site follow-up visits at 1-, 3-, and 6-months following subject's last (30th) treatment session.

DETAILED DESCRIPTION:
Screening procedures:

Prospective participants will be recruited for participation and informed consent will be obtained after all information is presented and all questions are answered to the patient's satisfaction. Once informed consent is obtained, the study team will confirm the patient meets all inclusion criteria and no exclusion criteria.

The following is a list of all assessments and tests that are required during the screening visit.

* Medical history, demographics, and Rutherford Class, vital signs, & circumference measurement of one calf.
* Ankle Brachial Index and Toe Brachial Index (ABI/TBI) will be measured at screening to determine eligibility and baseline values.
* Ultrasonography and Perfusion Imaging of the Foot will be undertaken prior to, during and after application of the VibratoSleeve TUS. All patients will undergo arterial duplex ultrasound at the level of the calf, ankle and/or foot to document the baseline vessel diameter, vessel velocity and volume flow. Perfusion imaging of the foot will be completed, using non-invasive methods like Flowmet by Medtronic, Inc. and Clarifi system by Modulim.

Treatments:

The initial three VibratoSleeve therapy sessions in this study will be performed at a clinical research center (VISOC).

Only subjects who have met all the inclusion criteria and none of the exclusion criteria will receive therapy. The device will be fitted and operated by Vibrato team member(s) while accompanied by site study staff. Study-related imaging will be performed by licensed vascular ultrasound technicians.

After pre-treatment imaging, Vibrato staff will fit the device to the posterior calf and couple it to skin with ultrasound gel. Therapy will be initiated using a Vibrato generator, gradually increasing acoustic output over the first 5 minutes of therapy to a nominal goal peak negative pressure, while assessing patient comfort.

During the first three 90-minute therapy sessions, ABI, TBI, ultrasonography and perfusion imaging of foot will be performed pre-treatment, during the 90-minute treatment, and immediately after the end of treatment, using identical methods to those described for screening (see above). It should be noted that ultrasound administration can be immediately stopped at any point in the 90-minute treatment period if there is significant subject discomfort or any evidence of an adverse event. Adverse events (if any) will also be recorded and assessed.

After the treatment measurements are completed, each subject will be asked to complete a questionnaire to capture subject's therapeutic experience. The feedback obtained may be used in developing future design enhancements of the VibratoSleeve device and/or a future pivotal trial design.

After the first three of 30 scheduled therapy sessions are completed, 25 of the remaining 27 sessions may be done at either the clinic or the patient's home, based upon subject's convenience and preference. A Vibrato representative will be present for all treatments to ensure proper operation and protocol compliance. No diagnostic/perfusion measurements will be taken during at-home sessions.

A mid-treatment session (number 15 +/- 2 sessions) and the last session (number 30) will be done in identical manner to the first treatment in the clinic, including all the perfusion measurements. After the final 30th treatment, subjects will commit to 1-, 3-, and 6-month follow up visits to assess the durability of the treatment.

All 30 treatments will be done within 45 days to allow subjects the option of receiving treatments 5 days per week, over a 6-week time frame.

One-, three- and six-month follow up visits:

At each follow-up visit, the subject will receive the same diagnostic and perfusion measurements as carried out during treatment sessions:

* ABI/TBI
* Ultrasonography at calf level
* Perfusion Imaging of foot
* Adverse events (if any) will also be identified, recorded and assessed, not only for clinic visits but also for at-home treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥22
2. Diagnosis of infrapopliteal PAD.
3. Rutherford class 3, 4 or 5 as determined by the investigator.
4. Toe Brachial Index (TBI) ≤ 0.6 OR Toe Blood Pressure ≤ 50 mmHg.

Exclusion Criteria:

1. Prior stenting in posterior tibial, anterior tibial or peroneal artery.
2. Re-vascularization procedure within 25 days prior to enrollment in the study. (Note: Patients who had re-vascularization procedure earlier than 25 days prior to enrollment are eligible for enrollment if all other criteria are met).
3. Ulcers, cellulitis, or skin breakdown in treatment areas (posterior calf).
4. History or diagnosis of severe chronic venous insufficiency or mixed arterio-venous disease.
5. Acute limb ischemia within 30 days prior to treatment.
6. History or diagnosis of deep venous thrombosis below the knee in treatment leg.
7. Uncontrolled diabetes defined as HbA1c greater than 10%.
8. Any conditions that, in the opinion of the investigator, may render the patient unable to complete the study or lead to difficulties for patient compliance with study requirements, or could confound study data.
9. Patient's enrollment in another investigational study that has not completed the required primary endpoint follow-up period (Note: Patients involved in a long-term surveillance phase of another study are eligible for enrollment in this study).

Eligibility for patients with bi-lateral PAD will be assessed based on the leg that has more advanced PAD. For bi-lateral PAD patients only one leg with the more advanced bi-lateral PAD will be treated.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-01-14 (Actual); Primary Completion 2023-02-10 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Changes in foot perfusion | Through study completion, an average of 6 months
  (2) Mean difference between pre-treatment (baseline) and post-treatment, and at the 1-, 3-, and 6-months post-treatment follow up visits, using Clarifi Imaging System (Modulim), which uses spatial frequency domain imaging (SFDI), to measure tissue oxygen saturation (StO2) and tissue hemoglobin (Hb) in the dermal microcirculation (HbT1) and macrocirculation (HbT2) to assess lower extremity blood supply.

SECONDARY OUTCOMES:
Subject Questionnaire | Through study completion, an average of 6 months.
  Based upon subject's perceptions during treatment sessions
Adverse Events | Through study completion, an average of 6 months.
  Analysis of all reported adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Vascular & Interventional Specialists of Orange County, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No
Data summaries and study conclusions will be shared with other researchers. Individual participant data will be unshared.

REFERENCES:
- [Result] Nazer B, Ghahghaie F, Kashima R, Khokhlova T, Perez C, Crum L, Matula T, Hata A. Therapeutic Ultrasound Promotes Reperfusion and Angiogenesis in a Rat Model of Peripheral Arterial Disease. Circ J. 2015;79(9):2043-9. doi: 10.1253/circj.CJ-15-0366. Epub 2015 Jun 9. PMID 26062950